CLINICAL TRIAL: NCT03586999
Title: Nivolumab With Standard of Care Chemotherapy for the First Line Treatment of Peripheral T Cell Lymphoma
Brief Title: Nivolumab With Standard of Care Chemotherapy for Peripheral T Cell Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0708.cc
Record Dates: First submitted 2018-06-29; First posted 2018-07-16 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Nivolumab; First Line Treatment; EPOCH; Standard of Care
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Nivolumab; Etoposide; Prednisolone; prednisolone phosphate; Methylprednisolone; Vincristine; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and EPOCH (Experimental): Patients will all receive nivolumab in combination with standard dose adjusted EPOCH for a planned 6 cycles, unless treatment is stopped early for disease progression or toxicity. Patients that have already received up to 1 cycle of standard of care chemotherapy will receive 5 cycles of experimental nivolumab + DA-EPOCH (dose adjusted, continuous infusion etoposide, prednisone, vincristine, doxorubicin, and bolus dosing of cyclophosphamide) for a total of 6 cycles of chemotherapy.
  Interventions: Drug: Nivolumab; Drug: Etoposide; Drug: Prednisolone; Drug: Oncovin; Drug: Cyclophosphamide; Drug: Hydroxydaunorubicin

INTERVENTIONS:
Drug: Nivolumab — Nivolumab injection is to be administered as an IV infusion.
  Other Names: Opdivo
Drug: Etoposide — Dosage calculations will be based on the patient's body surface area (BSA) at baseline, recommend using the Mosteller formula and administered through IV. Dose adjustments at the beginning of each cycle do not need to be made unless there has been a >10% weight gain or loss. Patients receive six 21-day cycles of the medications.
  Other Names: Vepesid; Toposar
Drug: Prednisolone — Dosage calculations will be based on the patient's body surface area (BSA) at baseline, recommend using the Mosteller formula and administered through IV. Dose adjustments at the beginning of each cycle do not need to be made unless there has been a >10% weight gain or loss. Patients receive six 21-day cycles of the medications.
  Other Names: Oraped; PediaPred; Millipred
Drug: Oncovin — Dosage calculations will be based on the patient's body surface area (BSA) at baseline, recommend using the Mosteller formula and administered through IV. Dose adjustments at the beginning of each cycle do not need to be made unless there has been a >10% weight gain or loss. Patients receive six 21-day cycles of the medications.
  Other Names: Vincristine; Leurocristine
Drug: Cyclophosphamide — Dosage calculations will be based on the patient's body surface area (BSA) at baseline, recommend using the Mosteller formula and administered through IV. Dose adjustments at the beginning of each cycle do not need to be made unless there has been a >10% weight gain or loss. Patients receive six 21-day cycles of the medications.
  Other Names: cytophosphane
Drug: Hydroxydaunorubicin — Dosage calculations will be based on the patient's body surface area (BSA) at baseline, recommend using the Mosteller formula and administered through IV. Dose adjustments at the beginning of each cycle do not need to be made unless there has been a >10% weight gain or loss. Patients receive six 21-day cycles of the medications.
  Other Names: Adriamycin

SUMMARY:
This regimen aims to become the first line treatment for peripheral T cell lymphoma, using nivolumab with the standard of care chemotherapy.

DETAILED DESCRIPTION:
Patients in this study will receive nivolumab in combination with the standard of care dose-adjusted EPOCH (etoposide, prednisone, vincristine, doxorubicin, cyclophosphamide) for six 21 day cycles. Patients will then have an autologous stem cell transplant or continue to receive maintenance therapy with nivolumab.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be a male or female aged 18-80.
4. Histologically confirmed new diagnosis of Stage II, III or IV Peripheral T-cell Non-Hodgkin's lymphoma not otherwise specified (NOS), Anaplastic large cell lymphoma (ALK-negative) (ALK-positive if IPI 3, 4, or 5), Angioimmunoblastic T-cell lymphoma, Enteropathy associated T-cell lymphoma (MEITL and EATL), Hepatosplenic T-cell lymphoma, y/8 T-cell lymphoma, Subcutaneous panniculitis-like T-cell lymphoma, and Nodal T-cell lymphomas with T-follicular helper phenotype.
5. Available pathology material (fine needle aspirate is inadequate) for review at the University of Colorado.
6. No prior therapy with the exception of prior radiation therapy and/or 1 cycle of chemotherapy (may be any chemotherapy regimen or even prednisone alone) based on current diagnosis and clinical condition. If given cytotoxic chemotherapy (one cycle only, e.g. CHOP), this cycle of treatment will count toward the 6 cycles of treatment given in the study.
7. ECOG performance status 0 - 2.
8. Laboratory status as follows:

   * ANC > 1000 cells/mm3, unless cytopenias due to lymphoma (i.e., bone marrow involvement or splenomegaly)
   * Platelet Count > 100,000 /μL, or > 50,000 /μL if bone marrow involvement or splenomegaly
   * Total bilirubin ≤1.5 x upper normal limit, or ≤ 3 x upper normal limit if documented hepatic involvement with lymphoma, or ≤ 5 x upper normal limit if history of Gilbert's Disease.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper normal limit (≤ 5 x upper normal limit if documented hepatic involvement with lymphoma).
   * Serum creatinine < 2.0 mg/dL or calculated creatinine clearance (CrCl) > 45 mL/min (Cockcroft-Gault, Appendix)
   * PT or INR, and PTT ≤ 1.5 x upper limit of normal unless patient is receiving anticoagulants. If patient is on warfarin therapy, levels should be within therapeutic range.
9. Patients with measurable disease. Measurable disease is defined as having at least one objective measurable disease parameter. A clearly defined, bi-dimensionally measurable defect or mass measuring at least 1.5 cm in diameter on the CT portion of a PET/CT or CT scan or MRI (if appropriate) will constitute measurable disease. Proof of lymphoma in the liver is required by a confirmation biopsy unless there is measurable disease by imaging. Skin lesions can be used as measurable disease provided bi-dimensional measurements are possible. Patients with non-measurable but evaluable disease may be eligible after discussion with the PI. Abnormal PET/CT scans will not constitute evaluable disease, unless verified by the CT scan portion, CT scan, or other appropriate imaging.
10. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use of contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 180 days after the last study treatment. A woman is considered to be of childbearing potential if she is post-menarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
11. Patient must be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. An additional malignancy treated with palliative intent within the past 2 years. Malignancies in patients who have completed definitive treatment with curative intent >1 year will be permitted after discussion with the PI. Adequately treated basal cell, squamous cell skin cancer, or thyroid cancer; carcinoma in situ of the cervix or breast; prostate cancer of Gleason Grade 6 or less with stable PSA levels are allowed.
2. Patients with a diagnosis of other PTCL histologies other than those specified in the inclusion criteria.
3. Primary T-cell CNS lymphoma; however, secondary CNS disease is not an exclusion criteria.
4. Pregnant or breastfeeding females.
5. Contraindication to any of the required concomitant drugs or supportive treatments.
6. Any other clinically significant medical disease or condition laboratory abnormality or psychiatric illness that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.
7. Ejection fraction of <45% by either MUGA or ECHO.
8. Has immunodeficiency or is being treated with immuno-suppressive therapy (aside from medications used to treat lymphoma) within 7 days of first dose of study treatment. Inhaled or topical steroids are accepted. Prednisone used to treat adrenal insufficiency in the absence of auto-immune disease is also acceptable.
9. Auto-immune condition requiring immuno-suppressive disease modifying therapy within the prior 2 years. Replacement therapy, e.g. levothyroxine for thyroiditis or insulin for diabetes are acceptable.
10. History of non-infectious pneumonitis requiring immuno-suppressive therapy.
11. Active hepatitis B or C (with measurable virus or antigen in serum) or HIV. Patients who are seropositive because of hepatitis B virus vaccine or have a history of hepatitis B (with no measurable virus or antigen in serum) are eligible.
12. Prior PD-1 or PD-L1 antibody treatment.
13. Has received a live virus vaccine in 30 days preceding start of therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Haverkos, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - City of Hope Cancer Center, Duarte, California
  - University of Colorado Hospital, Aurora, Colorado
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmitz N, Trumper L, Ziepert M, Nickelsen M, Ho AD, Metzner B, Peter N, Loeffler M, Rosenwald A, Pfreundschuh M. Treatment and prognosis of mature T-cell and NK-cell lymphoma: an analysis of patients with T-cell lymphoma treated in studies of the German High-Grade Non-Hodgkin Lymphoma Study Group. Blood. 2010 Nov 4;116(18):3418-25. doi: 10.1182/blood-2010-02-270785. Epub 2010 Jul 21. PMID 20660290
- [Background] Vose J, Armitage J, Weisenburger D; International T-Cell Lymphoma Project. International peripheral T-cell and natural killer/T-cell lymphoma study: pathology findings and clinical outcomes. J Clin Oncol. 2008 Sep 1;26(25):4124-30. doi: 10.1200/JCO.2008.16.4558. Epub 2008 Jul 14. PMID 18626005
- [Background] Ellin F, Landstrom J, Jerkeman M, Relander T. Real-world data on prognostic factors and treatment in peripheral T-cell lymphomas: a study from the Swedish Lymphoma Registry. Blood. 2014 Sep 4;124(10):1570-7. doi: 10.1182/blood-2014-04-573089. Epub 2014 Jul 8. PMID 25006130
- [Background] Maeda Y, Nishimori H, Yoshida I, Hiramatsu Y, Uno M, Masaki Y, Sunami K, Masunari T, Nawa Y, Yamane H, Gomyo H, Takahashi T, Yano T, Matsuo K, Ohshima K, Nakamura S, Yoshino T, Tanimoto M. Dose-adjusted EPOCH chemotherapy for untreated peripheral T-cell lymphomas: a multicenter phase II trial of West-JHOG PTCL0707. Haematologica. 2017 Dec;102(12):2097-2103. doi: 10.3324/haematol.2017.167742. Epub 2017 Sep 29. PMID 28971899
- [Background] Dunleavy K, Pittaluga S, Shovlin M, Roschewski M, Lai C, Steinberg SM, Jaffe ES, Wilson WH. Phase II trial of dose-adjusted EPOCH in untreated systemic anaplastic large cell lymphoma. Haematologica. 2016 Jan;101(1):e27-9. doi: 10.3324/haematol.2015.131151. Epub 2015 Oct 30. No abstract available. PMID 26518748
- [Background] Ghafouri S, Fenerty K, Schiller G, de Vos S, Eradat H, Timmerman J, Larson S, Mead M. Real-World Experience of Axicabtagene Ciloleucel and Tisagenlecleucel for Relapsed or Refractory Aggressive B-cell Lymphomas: A Single-Institution Experience. Clin Lymphoma Myeloma Leuk. 2021 Dec;21(12):861-872. doi: 10.1016/j.clml.2021.07.002. Epub 2021 Jul 19. PMID 34389271

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab and EPOCH
Started | 18
Completed | 16
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab and EPOCH
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.16 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Complete Response Rate
Description: Efficacy will be measured according to 2017 RECIL criteria. Responses will be assessed by the investigator and will be based on PET/CT scan to be obtained after 6 cycles of induction chemotherapy.
Time Frame: up to 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and EPOCH
Number analyzed (Participants) | 18
Participants | 11
Statistical Analysis 1: Comparison: Nivolumab and EPOCH; The study was to be suspended, if, at any time, there was sufficient evidence to suggest that the true probability of achieving a complete response falls below 30% while assuming the treatment drug will elicit a 56% complete response rate. Statistically significant evidence for this low complete response rate is defined as an observed complete response rate whose upper one-sided 90% confidence limit is 0-30%. Sample size calculations were made assuming 80% power; Test type: Superiority; p = .1, t-test, 2 sided — The proportion achieving a complete response will be calculated and will compared to null proportion of 30%. The population proportion for complete response rate, p-value and 90% confidence intervals for the complete response rate will be calculated; proportion = 0.3

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Toxicity analysis of nivolumab will be summarized by dose and severity as assessed by the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0 and relationship to study drug or the amount of grade 4-5 non-hematologic toxicities.
Time Frame: up to 100 days after last dose of nivolumab
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and EPOCH
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Efficacy: Overall Response Rate
Description: Efficacy will be measured according to 2017 RECIL criteria. Responses will be assessed by the investigator and will be based on PET/CT scan to be obtained after 6 cycles of induction chemotherapy. Complete response (CR), complete disappearance of all target lesions and Deauville score 1-3. Partial response (PR), ≥30% decrease in the sum of longest diameters of target lesions but not a CR and Deauville score 4-5. Stable disease (SD), <30% decrease or ≤ 20% increase in the sum of longest diameters of target lesions. Progressive disease (PD), >20% increase in the sum of longest diameters of target lesions, For small lymph nodes measuring < 15 mm post-therapy, a minimum of 5 mm increase in longest diameter to > 15 mm, or new lesions.
Time Frame: up to 100 days post transplant
Population: All patients on trial.
Measure: Count of Participants; unit: Participants
Groups:
- Nivo and EPOCH: Patients will all receive nivolumab in combination with standard dose adjusted EPOCH for a planned 6 cycles, unless treatment is stopped early for disease progression or toxicity. Patients that have already received up to 1 cycle of standard of care chemotherapy will receive 5 cycles of experimental nivolumab + DA-EPOCH (dose adjusted, continuous infusion etoposide, prednisone, vincristine, doxorubicin, and bolus dosing of cyclophosphamide) for a total of 6 cycles of chemotherapy.
Arm/Group | Nivo and EPOCH
Number analyzed (Participants) | 18
Participants | 16

4. Secondary Outcome: Efficacy: Progression Free Survival Rate
Description: as for outcome 1
Time Frame: up to 2 years after completion of treatment
Population: All patients treated on trial.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivo and EPOCH
Number analyzed (Participants) | 18
months | 14.5 [7.5 to 22.2]

5. Secondary Outcome: Efficacy: Event Free Survival
Description: Efficacy will be measured according to 2017 RECIL criteria. Responses will be assessed by the investigator and will be based on PET/CT scan to be obtained after 6 cycles of induction chemotherapy. Events defined as start of new treatment, progression, or death.
Time Frame: up to 2 years after completion of treatment
Population: All patients treated on trial
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivo and EPOCH
Number analyzed (Participants) | 18
months | 10.5 [6.9 to 20.5]

6. Secondary Outcome: Immune-related Predictors of Response
Description: We assessed PD-L1 expression using immunohistochemistry on pre-treatment tumor tissue. The outcome of measurement was complete response yes vs. no. Using logistic regression, we assessed if the percentage of PDL1+ cells was predictive of achieving a complete response.
Time Frame: Within 6 months of treatment
Population: Only 17 participants had tumor tissue available.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Nivo and EPOCH
Number analyzed (Participants) | 17
odds ratio | 0.985 [0.938 to 1.034]

ADVERSE EVENTS:
Time Frame: up to 100 days after last dose of nivolumab
Arm/Group | Nivolumab and EPOCH
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 13/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and EPOCH (N=18)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Fever (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
chest wall pain (Cardiac disorders) | 1 (1)
iliacus/iliopsoas hematoma (Injury, poisoning and procedural complications) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 1 (1)
Clostridioides difficile (Gastrointestinal disorders) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Chemotherapy Extravasation (Injury, poisoning and procedural complications) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
dermatologic toxicity c/w Stevens Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Elevated Transaminases (Blood and lymphatic system disorders) | 1 (1)
intra-abdominal infection (Infections and infestations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Infected Biopsy Site (Infections and infestations) | 1 (1)
neutropenic fever c/f SIRS (Infections and infestations) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sepsis (Infections and infestations) | 3 (4)
Syncopal Episodes (Psychiatric disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and EPOCH (N=18)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Abdominal soft tissue nodules (General disorders) | 1 (1)
Abnormal Coordination (General disorders) | 1 (1)
activity change (General disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
acute skin pain 2/2 dermatologic toxicity (Skin and subcutaneous tissue disorders) | 1 (1)
Acute tailbone (coccyx) pain (Injury, poisoning and procedural complications) | 2 (4)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4)
Alkaline phosphatase increased (Investigations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 7 (23)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
asymptomatic bradycardia (intermittent) (Cardiac disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
autoimmune thyroiditis (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Bacteremia (Infections and infestations) | 1 (1)
benign prostatic hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
biapical predominant ground glass opacities - chest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
bilateral nephrolithiasis (Renal and urinary disorders) | 1 (1)
bilateral pneumonic infiltrates (Infections and infestations) | 1 (1)
bladder spasms (Renal and urinary disorders) | 1 (1)
blisters to feet c/w SJS (General disorders) | 1 (1)
blisters to palms c/w SJS (General disorders) | 1 (1)
blood bilirubin increased (Investigations) | 2 (2)
Elevated systolic blood pressure (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 3 (4)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
chest pain (Cardiac disorders) | 2 (2)
Chills (General disorders) | 7 (9)
chronic hypercapnic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
chronic pain syndrome (General disorders) | 1 (1)
Chronic venous stasis (General disorders) | 1 (1)
erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Concentration impairment (General disorders) | 2 (2)
Confusion (Psychiatric disorders) | 5 (6)
Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 9 (11)
costovertebral angle pain - left (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
COVID-19 (Infections and infestations) | 1 (1)
deconditioning (Musculoskeletal and connective tissue disorders) | 1 (1)
decreased calorie intake (Metabolism and nutrition disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
dermatologic toxicity c/w Stevens Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (13)
Disseminated intravascular coagulation (Vascular disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (8)
Dry eye (Eye disorders) | 3 (3)
Dry mouth (General disorders) | 1 (1)
Dry nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
dyslipidemia (Metabolism and nutrition disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
dystonia (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
ECOG increase (General disorders) | 1 (1)
Edema (General disorders) | 10 (22)
elevated lactate (General disorders) | 2 (3)
elevated LDH (intermittent) (Blood and lymphatic system disorders) | 1 (1)
Elevated PSA (General disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (7)
Fatigue (General disorders) | 8 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Fever (General disorders) | 8 (12)
Fluid Overload (General disorders) | 3 (3)
Foot Drop (Nervous system disorders) | 1 (1)
frequent urination (Renal and urinary disorders) | 1 (1)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 2 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
gum oozing and bleeding (General disorders) | 1 (1)
gum soreness (General disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 2 (2)
Headache (General disorders) | 7 (8)
heart failure with preserved ejection fraction (Cardiac disorders) | 1 (1)
Hematuria (Blood and lymphatic system disorders) | 2 (2)
Hemophagocytic lymphohistiocytosis (HLH) (Blood and lymphatic system disorders) | 1 (1)
Hemrrohoids (General disorders) | 1 (1)
Hiccups (General disorders) | 1 (1)
enteritis (Infections and infestations) | 1 (1)
Hoarseness (General disorders) | 2 (2)
Hot flashes (Reproductive system and breast disorders) | 2 (2)
hyperbilirubinemia (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (8)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 6 (21)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (15)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (9)
hypotension (Vascular disorders) | 4 (9)
Hypothyroidism (Endocrine disorders) | 3 (3)
hypovolemia (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (8)
hypervolemia (Vascular disorders) | 3 (3)
immunocompromised (General disorders) | 1 (1)
non st elevation myocardial infarction (NSTEMI) (Cardiac disorders) | 1 (1)
influenza A (General disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
right side tongue sore (Skin and subcutaneous tissue disorders) | 1 (1)
rigors (Musculoskeletal and connective tissue disorders) | 1 (1)
sensory deficit (Nervous system disorders) | 1 (1)
left-sided parasthesia in groin area (Musculoskeletal and connective tissue disorders) | 1 (1)
Lesion (Skin and subcutaneous tissue disorders) | 3 (4)
Lethargy (Nervous system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 5 (6)
Liver Injury (Injury, poisoning and procedural complications) | 1 (1)
low absolute lymphocyte (Blood and lymphatic system disorders) | 2 (4)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
maxillary sinus nodular mucosal thickening (Skin and subcutaneous tissue disorders) | 1 (1)
Memory impairment (Psychiatric disorders) | 1 (1)
Methicillin-resistant Staphylococcus aureus (MRSA) (Infections and infestations) | 1 (1)
mouth sore (Skin and subcutaneous tissue disorders) | 2 (2)
Mucositis (Skin and subcutaneous tissue disorders) | 5 (8)
multifocal infection of the lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
small bilateral pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (12)
Neuralgia (Nervous system disorders) | 1 (1)
neuropathy (Nervous system disorders) | 11 (22)
Neutrophil count decreased (Investigations) | 1 (8)
oral aphthous ulcerations (Skin and subcutaneous tissue disorders) | 1 (1)
oral candidiasis (Infections and infestations) | 2 (2)
Pain (General disorders) | 9 (18)
parenchymal lung abnormality (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 2 (14)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
posterior oropharyngeal erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (7)
Retroperitoneal hemorrhage (Eye disorders) | 1 (1)
rhinovirus (Infections and infestations) | 1 (1)
right parotid mass with slight drainage and erythema (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 6 (7)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Skin Sloughing (Skin and subcutaneous tissue disorders) | 1 (2)
small bowel ileus (Gastrointestinal disorders) | 1 (1)
small lump on right wrist (General disorders) | 1 (1)
Sore throat (General disorders) | 3 (4)
splenic artery thrombosis (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Syndrome of inappropriate antidiuretic hormone secretion (SIADH) (General disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
throat tightening (General disorders) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Transaminitis (Gastrointestinal disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
uretal stone (Renal and urinary disorders) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 2 (3)
urolithiasis (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
weakness (General disorders) | 6 (9)
Weight loss (Metabolism and nutrition disorders) | 3 (3)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (3)
wrist dislocation (Musculoskeletal and connective tissue disorders) | 1 (1)
tenderness (Skin and subcutaneous tissue disorders) | 2 (2)
Unstable balance (Nervous system disorders) | 1 (1)
watering eyes (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03586999/Prot_SAP_ICF_000.pdf